CLINICAL TRIAL: NCT06948071
Title: Enhanced Recovery Protocol for Acute, Complicated Appendicitis After Laparoscopic Appendectomy: An Exploratory Pilot Study
Brief Title: Enhanced Recovery After Surgery (ERAS) for Complicated Appendicitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Galinos Barmparas, MD, Staff Physician II, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003804
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Appendicitis Acute; Appendicitis Perforated; Appendicitis With Perforation; Appendicitis Suppurative; Appendicitis Gangrenous
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ERAS (Other): Patients with intraoperative diagnosis of complicated appendicitis as determined by the operating surgeon.
  Interventions: Other: Discharge on oral antibiotics

INTERVENTIONS:
Other: Discharge on oral antibiotics — Patients will be discharged to home on an oral antibiotic regimen for 3 days instead of being admitted for intravenous antibiotics.

SUMMARY:
The exploratory objective of this pilot study is to evaluate the feasibility and safety of an enhanced recovery protocol that will allow adult patients to be discharged to home on an oral antibiotic regimen for three days following a laparoscopic appendectomy for complicated appendicitis. Feasibility will be determined by high compliance and adherence of patients to the postoperative instructions, while safety will be assessed by the incidence of postoperative infectious complications and requirement for re-admission.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18 and 65 years of age.
* Patients undergoing a laparoscopic appendectomy.
* Diagnosis of complicated appendicitis based on pre-operative imaging or intra-operative assessment. The definition of a complicated appendicitis will include: (a) perforated appendicitis, without generalized peritonitis; (b) gangrenous appendicitis, without generalized peritonitis; (c) suppurative appendicitis; (d) iatrogenic perforation of the appendix.
* Meet criteria for discharge from the post-anesthesia care unit (PACU).
* Ability to reliably follow up with the study procedures.

Exclusion Criteria:

* Age < 18 years or > 65 years.
* Pregnancy.
* Homelessness.
* Patients who present with generalized peritonitis.
* Patients with comorbid conditions, including diabetes mellitus, immunosuppressed state for any reason, patients on chronic anticoagulation (excluding Aspirin 81 mg).
* Patients who present with septic shock.
* Patients who require conversion to an open appendectomy.
* Patients who present with additional findings on imaging studies or intra-operatively, including ileus or small bowel obstruction.
* Based on surgeon's clinical judgment for reasons that may not be outlined above.
* Allergy or intolerance to study medication(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-21 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Readmission rate | 30 days
  Feasibility will be determined by the readmission within 30 days rate for any reason
Postoperative infections | 30 days
  Safety will be assessed by the incidence of postoperative infectious complications

CONTACTS AND LOCATIONS:
Overall Officials: Galinos Barmparas, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van Rossem CC, Schreinemacher MH, van Geloven AA, Bemelman WA; Snapshot Appendicitis Collaborative Study Group. Antibiotic Duration After Laparoscopic Appendectomy for Acute Complicated Appendicitis. JAMA Surg. 2016 Apr;151(4):323-9. doi: 10.1001/jamasurg.2015.4236. PMID 26580850
- [Background] van den Boom AL, de Wijkerslooth EML, Giesen LJX, van Rossem CC, Toorenvliet BR, Wijnhoven BPL. Postoperative Antibiotics and Time to Reach Discharge Criteria after Appendectomy for Complex Appendicitis. Dig Surg. 2022;39(4):162-168. doi: 10.1159/000526790. Epub 2022 Aug 30. PMID 36041400
- [Background] Kleif J, Rasmussen L, Fonnes S, Tibaek P, Daoud A, Lund H, Gogenur I. Enteral Antibiotics are Non-inferior to Intravenous Antibiotics After Complicated Appendicitis in Adults: A Retrospective Multicentre Non-inferiority Study. World J Surg. 2017 Nov;41(11):2706-2714. doi: 10.1007/s00268-017-4076-6. PMID 28600695
- See also: Postoperative antibiotic therapy after appendectomy in patients with non-perforated appendicitis - PMC. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5494044/